CLINICAL TRIAL: NCT02672384
Title: Chronic Periodontitis in Critically Ill Patients: Diagnosis and Epidemiology
Acronym: CP-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-ICU STUDY (RB 15.108)
Record Dates: First submitted 2015-09-18; First posted 2016-02-03 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Chronic Periodontitis; Intensive Care Unit
Keywords: Intensive care unit; Invasive mechanical ventilation; Chronic periodontitis; Point of Care P. gingivalis test
MeSH Terms: conditions — Chronic Periodontitis | interventions — Diagnosis, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients in ICU (Experimental): Dental examination will be performed to diagnose CP based on the Centre for Diseases Control definition.
  A point of care P. gingivalis test (Denka Seiken Co (Japan) ) on saliva and detection of antibodies against P. gingivalis in sera will be performed.
  In case of discrepancies between both diagnoses methods, RT-PCR for identification of P. gingivalis and other pathogens will be performed on samples of periodontal pocket performed in routine.
  Interventions: Procedure: Dental examination and a point of care P. gingivalis test (Denka Seiken Co (Japan) )

INTERVENTIONS:
Procedure: Dental examination and a point of care P. gingivalis test (Denka Seiken Co (Japan) ) — Dental examination Study exams (oral and blood sample collection)

SUMMARY:
This study evaluates the diagnostic performances of Point of Care P. gingivalis test in saliva with serum IgG P. gingivalis, in reference to dental examination as a gold standard in patients hospitalised in intensive care unit (ICU)

DETAILED DESCRIPTION:
Chronic Periodontitis (CP) is a common but under diagnosed chronic infection and inflammation of the periodontal tissue. Porphyromonas gingivalis is one of the most common pathogens associated with CP. In patients hospitalised in Intensive Care Unit (ICU), P. gingivalis has been reported to be associated with Ventilator-Associated Pneumonia (VAP).

This pilot study evaluate an easily accessible method the Point of care P. gingivalis tests on saliva and detection of antibodies against P. gingivalis in sera (already validated to diagnose CP in the general population) to dental examination as a gold standard, in ICU patients.

A biobank from critically ill patients will be establish for future oral health research in this patient population: for about 50 patients with both samples available, at enrolment and at day 5 +/-2 days after enrolment. Oral pathogens of different sites (tongue, saliva, dental plaque, internal jaw) at enrolment and at day 5 +/- 2 days after enrolment. Samples of periodontal pocket will be collected only for patients diagnosed with CP. When patients will have a pulmonary sample performed in routine, pulmonary sample will also be stored. Plasma and sera will also be taken at enrolment and stored for further research on P. gingivalis and inflammation in ICU patients Patients will be enrolled and will be contacted after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Admitted to medical or surgical intensive care unit
* Invasive mechanical ventilation for an anticipated duration of at least 48 hours

Exclusion Criteria:

* Edentulous
* Known to be pregnant
* ICU stay<48 hours
* High risk of infectious endocarditis
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Result (positive/negative) of the point-of-care P. gingivalis test in saliva and P. gingivalis antibodies in sera | one day
  P. gingivalis test in saliva and P. gingivalis antibodies in sera

SECONDARY OUTCOMES:
Ratio of enrolled patients/eligible patients | one year
  compare listing of enrolled patients and eligible patients
Number of patient with discrepancies in findings of dental exam and point of care P. gingivalis test combined | 90 days
  measure of discrepancies in findings of dental exam and point of care P. gingivalis test combined
Mortality at 90 days after intubation | 90 days
  Mortality
Incidence of CP (Chronic periodontitis) in mechanically ventilated patients | 90 days
  CP (Chronic periodontitis) measure
Incidence of VAP(Ventilator-Associated Pneumonia) | 90 days
  VAP(Ventilator-Associated Pneumonia)
Recruitment rate | one year
  Recruitment rate

CONTACTS AND LOCATIONS:
Locations (1):
- Brest, University Hospital, Brest, France